CLINICAL TRIAL: NCT01203163
Title: Case Analysis on Real Life Incidence of PDT Safety Outcomes: Multicentre, Observational Post-marketing Safety Surveillance Registry of Patients Exposed to Photodynamic Therapy With Porfimer Sodium: The CALIPSO Registry
Brief Title: Case Analysis on Real Life Incidence of Photodynamic Therapy (PDT) Safety Outcomes
Acronym: CALIPSO
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor cancelled the study
Sponsor: Pinnacle Biologics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-PO-PHORC07-01
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Esophageal Cancer; Lung Cancer; Barrett's Esophagus
Keywords: PDT; porfimer sodium; esophageal cancer; NSCLC; HGD in BE
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms; Barrett Esophagus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PDT with porfimer sodium

SUMMARY:
Three main adverse reactions, namely photosensitivity (reaction that is similar to sunburn), oesophageal stenosis (narrowing or closure of the food pipe), perforation of the treated area (a tear or puncture of the tissue), have been identified in research studies evaluating photodynamic therapy (PDT) with porfimer sodium. Because of the low incidence of the disease or the variation in the occurrence of these adverse reactions among different indications, it is difficult to determine the occurrence and frequency of these safety issues in routine clinical practice.

This post-marketing safety surveillance registry is set-up to evaluate the safety of PDT using porfimer sodium. A registry allows the collection of data to evaluate real-world results in the practice of medicine. The registry will monitor the patient's health and any events, with a main focus on photosensitivity, oesophageal stenosis, and perforation of the treated area. This registry will involve 500 patients, across 20 to 36 hospitals in the US and Europe, scheduled to receive an injection of porfimer sodium with PDT for the treatment of lung cancer, esophageal [food pipe] cancer, or high-grade dysplasia (HGD) (precancerous change in the food pipe tissue) in Barrett's esophagus.

DETAILED DESCRIPTION:
Patients will be enrolled in the registry upon injection of the porfimer sodium. During normal medical examination, criteria for entry onto the registry will be verified to confirm eligibility, and medical procedures including demographic information, disease history, medical history, physical exam, and clinical laboratory testing performed under normal practice will be collected. Patients will receive PDT as per current practice and will be repeated as per the physician's judgment. All patients will be assessed as per current practice, that is usually at least three times, after a PDT session. Additional visits will be sought for those patients who are presenting photosensitivity reaction, esophageal stenosis, perforation at the site of laser light application, or any unresolved serious adverse reactions at the third visit after treatment. All patients will be requested by their physician to complete a two-part Daily Diary to record adverse reactions using a check-list form and a general section for reporting any adverse events and intake of concomitant medications at the time of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo PDT with Photofrin
* Patients must have the mental, literate, and legal ability to give a written informed consent, which must comply with the International Conference on Harmonization (ICH) guidelines and local requirements.

Exclusion Criteria:

* Patients treated with Photosan®
* Patients being treated with any investigational drug or participating in any interventional studies, with the exception of investigational photoprotection measures.
* Patients who are unable or unwilling to complete the follow-up evaluations required for the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from esophageal cancer, lung cancer, or HGD in Barrett's esophagus and scheduled to undergo PDT with porfimer sodium
Sampling Method: Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing Adverse Reactions of Special Interest | 3 months
  Proportion of patients experiencing photosensitivity reaction, oesophageal stenosis, and/or perforation at the site of laser light application after PDT.

SECONDARY OUTCOMES:
Incidence of the photosensitivity reaction in patients with liver insufficiency (disease) | 3 months
  Possible differences in the incidence of the photosensitivity reaction between patients with and without liver insufficiency
Relationships between photosensitivity reaction and skin color | 3 months
Overall safety in patients with renal insufficiency (disease) | 3 months